CLINICAL TRIAL: NCT06771232
Title: Impact of Lung Recruitment Maneuvers and Positive End-Expiratory Pressure (PEEP) on Intracranial Pressure in Patients Undergoing Cranial Surgery
Brief Title: Lung Recruitment and PEEP Effects on Intracranial Pressure in Cranial Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: OAIC 1463/24
Record Dates: First submitted 2024-12-11; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Pressure Increase; Mechanical Ventilation Complication
Keywords: Positive end expiratory pressure; intracranial pressure
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Subdural pressure measurement — Subdural intracranial pressure (SDIP) will observed during an alveolar recruitment maneuver and best PEEP titatration. SDIP will be measured while mechanical ventilation is maintained using the identified best PEEP.
  Other Names: Alveolar recruitment maneuver and decremental PEEP titration

SUMMARY:
High positive end-expiratory pressure (PEEP) levels required to achieve clinical benefits may increase ICP and reduce cerebral perfusion pressure (CPP) in patients at risk of intracranial hypertension.

However, individualizing ventilation parameters is essential for each patient. Among protective ventilation strategies, PEEP is key to preventing alveolar collapse. The PEEP level that minimizes alveolar collapse while avoiding overdistension of the pulmonary parenchyma is known as the Best PEEP. This study aims to evaluate the application of Best PEEP in cranial neurosurgery.

DETAILED DESCRIPTION:
In general anesthesia for neurosurgery, mechanical ventilation is the standard approach. However, mechanical ventilation can induce pulmonary parenchymal injury through various mechanisms, including volutrauma, barotrauma, and atelectrauma. These correspond to lung damage caused by high tidal volumes, elevated airway pressures, repetitive alveolar collapse, and reopening. Protective ventilation strategies include limiting tidal volume (Vt), applying positive end-expiratory pressure (PEEP), and performing alveolar recruitment maneuvers (ARM).

Historically, both ARM and higher levels of PEEP have been avoided in neurocritical patients, including those undergoing neurosurgery, due to concerns about their potential impact on intracranial pressure (ICP) and cerebral perfusion pressure (CPP). As postoperative pulmonary complications can significantly alter the prognosis of surgical patients, increasing hospital stay and healthcare costs, and, in neurocritical patients, compromising cerebral oxygenation, protective ventilation strategies may play a critical role in patients undergoing neurosurgery. Their historical exclusion from studies lacks demonstrated physiological justification.

Here, the investigators aim to evaluate the impact of intrathoracic pressure on ICP in neurosurgical patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-III.
* Elective cranial neurosurgery.

Exclusion Criteria:

* ASA classification IV or higher.
* Documented intracranial hypertension.
* Severe pulmonary disease (e.g., asthma, COPD).
* Emergency surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial disease undergoing elective intracranial surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Subdural intracranial pressure (sICP) mmHg | during the procedure
  Change in sICP during an alveolar recruitment maneuver (ARM)

SECONDARY OUTCOMES:
Pulmonary mechanics parameters | Intraoperative
  To describe pulmonary mechanics parameters, including plateau pressure (cmH2O) and driving pressure.(cmH2O)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Maldonado, M.D., M.Sc., Study Chair — Hospital Clinico de la Universidad de Chile
Locations (1):
- Hospital Clínico de la Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No